CLINICAL TRIAL: NCT06777342
Title: Effect of Preoperative Sleep Intervention on Postoperative Delirium in Adult Patients Undergoing Cardiac Surgery: a Multicenter Randomized Controlled Trial
Brief Title: Effect of Preoperative Sleep Intervention on Postoperative Delirium in Adult Patients Undergoing Cardiac Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yan Fuxia (Other)
Responsible Party: Sponsor-Investigator, Yan Fuxia, principal investigator, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-2417
Record Dates: First submitted 2025-01-06; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-11

CONDITIONS: Delirium - Postoperative; Sleep Problems; CABG; Valve Surgery
MeSH Terms: conditions — Emergence Delirium; Parasomnias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo group (Placebo Comparator)
  Interventions: Other: Placebo intervention
- Placebo and cognitive behavioral therapy intervention group (Experimental)
  Interventions: Behavioral: Cognitive behavioral therapy intervention; Other: Placebo intervention
- Melatonin and cognitive behavioral therapy intervention group (Experimental)
  Interventions: Behavioral: Cognitive behavioral therapy intervention; Dietary Supplement: Melatonin intervention

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy intervention — The cognitive behavioral intervention provides sleep-related education 7-14 days before surgery. The educational content should include the following aspects: 1) Establish a consistent bedtime and wake-up time, recommending a sleep schedule from 22:00 to 07:00, and avoid prolonged daytime naps; 2) Optimize the sleep environment by ensuring a quiet setting, turning off lights, and refraining from using mobile phones, computers, and other electronic devices 30 minutes before bedtime; 3) Manage diet by avoiding caffeinated foods such as chocolate, tea, and cola; 4) Engage in appropriate daytime activities as permitted by the patient's condition.
  Arms: Melatonin and cognitive behavioral therapy intervention group; Placebo and cognitive behavioral therapy intervention group
Dietary Supplement: Melatonin intervention — Patients in the melatonin intervention group are required to take an oral melatonin of 5 mg at 30-60 minutes before sleep (administered at 21:00) nightly for 7 to 14 days before surgery. The melatonin was provided by Kangenbei Pharmaceutical Co., LTD. (Hangzhou, Zhejiang, China).
  Arms: Melatonin and cognitive behavioral therapy intervention group
Other: Placebo intervention — Patients in the placebo group need to take oral placebos of 5 mg at 30-60 minutes (administered at 21:00) before sleep, nightly, for 7 to 14 days before surgery. The placebo is provided by Guangzhou Boji Biomedical Science Park Co., LTD. (Guangzhou, Guangdong, China).
  Arms: Placebo and cognitive behavioral therapy intervention group; Placebo group

SUMMARY:
This is a multicenter, randomized, controlled clinical trial aimed to determine whether preoperative sleep interventions could reduce the incidence of adverse outcomes, such as postoperative delirium, in adult patients undergoing cardiac surgery. The study will include adult patients undergoing coronary artery bypass grafting and/or valve surgery with concomitant sleep disorders, as assessed by the Pittsburgh Sleep Quality Index. All participants will be randomly assigned to placebo, placebo + cognitive behavioral therapy, and melatonin + cognitive behavioral therapy in a 1:1:1 ratio. The primary outcome is the incidence of postoperative delirium within 7 days after surgery or before discharge, and secondary outcomes include postoperative cognitive function, sleep quality, and severity and duration of delirium. The results of this study will provide suggestions for the prevention of delirium after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Scheduled for elective coronary artery bypass grafting and/or valve surgery.
3. Preoperative Pittsburgh Sleep Quality Index (PSQI) score ≥ 5.

Exclusion Criteria:

1. History of neurosurgery, cerebral hemorrhage, cerebral infarction, delirium, dementia, or other neurological diseases.
2. History of mental illness.
3. Habitual heavy drinking.
4. American Society of Anesthesiologists (ASA) grade IV or above.
5. Severe hepatic dysfunction (Child-Pugh Grade C) or renal dysfunction (chronic kidney disease stages 3-4).
6. Contraindications to melatonin use, such as allergies to melatonin-related ingredients.
7. Currently taking melatonin, melatonin receptor agonists, sleep-related medications, sedatives, antipsychotic medications, or opioids.
8. Inability to communicate due to hearing or speech impairment, or refusal to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1281 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative delirium | Postoperative 7 days or before discharge

SECONDARY OUTCOMES:
Postoperative sleep quality | Postoperative 7 days or before discharge
  The sleep quality was evaluated using the Actigraph model wGT3X-BT and the Sleep Quality and Nighttime Restlessness Scale (SQNRS) score. Subjects wore the Actigraph wGT3X-BT activity monitor from the beginning of their hospital admission until 7 days after surgery or before discharge. The device will record parameters such as total sleep time, wake time after falling asleep, number of awakenings, average wake time, and sleep efficiency during the first 7 days after surgery or before discharge to assess the subjects' sleep quality. Additionally, the SQNRS score was used to evaluate patients' subjective sleep quality during the same period. The SQNRS score ranges from 0 to 10, with higher scores indicating better sleep quality.
Postoperative cognitive function | The 7th day after surgery or before discharge
  The Montreal Cognitive Assessment (MoCA) will be administered to evaluate the cognitive function of the patients 7 days after surgery or before discharge. The MoCA has a total score of 30 points, with a score above 26 indicating normal cognitive function.
Duration and severity of delirium | Postoperative 7 days or before discharge
Postoperative mood and anxiety | The 7th day after surgery or before discharge
  The Hospital Anxiety and Depression Scale (HADS) will be utilized to evaluate the mood and anxiety levels of the patients during the first 7 days after surgery or before discharge. The HADS scale comprises two subscales, totalling 14 items: 7 items assess anxiety, and the other 7 assess depression. Each item is scored on a scale of 0 to 3, with each subscale totalling up to 21 points. Interpretation of the scores is as follows: 0-7 indicates a normal state, 8-10 suggests mild anxiety/depression, 11-14 indicates moderate anxiety/depression, and 15-21 suggests severe anxiety/depression.

OTHER OUTCOMES:
Postoperative pain score | Postoperative 7 days or before discharge
  The Visual Analogue Scale (VAS) will be employed to assess the pain levels of patients during the first 7 days after surgery or before discharge. A VAS score ranges from 0 to 10, with 1-3 indicating mild pain, 4-6 indicating moderate pain, and 7-10 indicating severe pain.
Types and doses of postoperative sedative and analgesic drugs | Postoperative 7 days or before discharge
Postoperative nausea and vomiting | Postoperative 7 days or before discharge
  The frequency of nausea and vomiting will be recorded daily for 7 days following surgery or before discharge, as documented during bedside consultations.
Postoperative markers of oxidative stress and inflammation | 24 hours after surgery
  Within 24 hours after surgery, levels of malondialdehyde (MDA), ascorbic acid (AA), dehydroascorbic acid (DHA), and C-reactive protein (CRP) will be determined from 5 mL of venous blood drawn from the patients.
Postoperative mechanical ventilation time and Intensive Care Unit stay time | Postoperative 7 days or before discharge
Length of hospital stay | 30 days after surgery
In-hospital mortality | Postoperative 7 days or before discharge
Serious adverse cardiovascular events | Postoperative 7 days or before discharge
Long-term survival | 30 days after surgery
  Survival information will be obtained through telephone follow-up.
Long-term survival | 12 months after surgery
  Survival information will be obtained through telephone follow-up.
Long-term sleep quality | 30 days after surgery
  The patients' sleep quality will be assessed through telephone follow-up using the Sleep Quality and Nighttime Restlessness Scale (SQNRS). The SQNRS score ranges from 0 to 10, with higher scores indicating better sleep quality.
Long-term sleep quality | 12 months after surgery
  The patients' sleep quality will be assessed through telephone follow-up using the Sleep Quality and Nighttime Restlessness Scale (SQNRS). The SQNRS score ranges from 0 to 10, with higher scores indicating better sleep quality.
Long-term pain | 30 days after surgery
  The patients' long-term pain will be assessed through telephone follow-up using the Visual Analogue Scale (VAS). A VAS score ranges from 0 to 10, with 1-3 indicating mild pain, 4-6 indicating moderate pain, and 7-10 indicating severe pain.
Long-term pain | 12 months after surgery
  The patients' long-term pain will be assessed through telephone follow-up using the Visual Analogue Scale (VAS). A VAS score ranges from 0 to 10, with 1-3 indicating mild pain, 4-6 indicating moderate pain, and 7-10 indicating severe pain.
Total hospitalization costs | 30 days after surgery

IPD SHARING:
Plan to Share IPD: No